CLINICAL TRIAL: NCT01962194
Title: Mapping and Stimulating the Limbic Areas of the Subthalamic Nucleus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE403-HMO-CTIL
Record Dates: First submitted 2013-09-25; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-06

CONDITIONS: Mapping the Limbic STN Using Neuronal Responses
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD and OCD paients for DBS intervention (Experimental): Parkinson's disease (PD; n=5) and obsessive-compulsive disorder (OCD; n=5) patients that are candidates for treatment with STN DBS will be recruited over a period of two years.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — In this study we will use implantable Deep Brain Stimulation (DBS) system with local field potential sensing capability. The Device is the Medtronic, Inc DBS Implantable System, "Activa PC+S", which has therapy equivalent to "Activa PC", and has a new sensing programmer.

SUMMARY:
The investigators hypothesize that the emotional and cognitive areas of the Subthalamic Nucleus (STN) have distinct electrophysiological properties and that specific stimulation of these areas can influence the mental and the emotional state. Parkinson's disease (PD; n=5) and obsessive-compulsive disorder (OCD; n=5) patients that are candidates for treatment with Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) will be recruited over a period of two years. The patients will be enrolled in a prospective, open label, clinical trial and will be followed for one year. No randomization or blinding will be used in this study.

ELIGIBILITY:
Inclusion criteria of PD patients:

1. Patients with PD who meet accepted criteria for DBS surgery:

   i. advanced idiopathic PD ii. long-term levodopa use that leads to decreased efficacy and increased incidence of adverse effects iii. normal cognitive function or mild-moderate cognitive decline (Addenbrooke's Cognitive Examination (ACE) > 75 and the Frontal Assessment Battery (FAB) > 10.
2. Age 40-75 years
3. Male or female
4. Competent and willing to give written informed consent

Exclusion Criteria of PD patients:

1. A diagnosis of severe major depression disorder (MDD) with psychotic features
2. Significant suicidal risk [Hamilton Depression scale item 3 (suicide) >2]
3. Lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months
4. Significant cognitive decline, as measured by Addenbrooke's Cognitive Examination (ACE) < 75 and the Frontal Assessment Battery (FAB) < 10.
5. Significant cognitive impairment that would affect a participant's ability to give informed consent or provide interview or self-report data reliably
6. Any clinically significant abnormality on preoperative MRI
7. Any DBS contraindication, infection, coagulopathy, significant cardiac risk factors, or other medical risk factors for surgery
8. Pregnant and/or woman of childbearing age not using effective forms of birth control

Inclusion criteria of OCD patients:

1. Obsessive-compulsive disorder (OCD), diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) (SCID-IV)
2. Presence of disabling severity, as assessed by a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 25
3. Documented highly treatment refractory OCD; the documentation must demonstrate persistence of severe symptoms and impairment for 5 or more years despite both pharmacological and psychological treatments.
4. Either drug free or on a stable drug regimen for at least 6 weeks before study entry
5. General good overall health
6. Age 20-70 years
7. Male or female
8. Competent and willing to give written informed consent.

Exclusion Criteria of OCD patients:

1. A diagnosis of severe major depression disorder (MDD) with psychotic features
2. Significant suicidal risk [Hamilton Depression scale item 3 (suicide) >2].
3. Comorbidity with any primary Psychotic Disorder, Bipolar Disorder, Post Traumatic Stress Disorder (PTSD), Eating Disorder.
4. Lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months
5. Significant cognitive decline, as measured by Addenbrooke's Cognitive Examination (ACE) < 75 and the Frontal Assessment Battery (FAB) < 10.
6. Significant cognitive impairment that would affect a participant's ability to give informed consent or provide interview or self-report data reliably
7. Any another current clinically significant neurological disorder or medical illness affecting brain function, other than a tic disorder
8. Any clinically significant abnormality on preoperative MRI
9. Any DBS contraindication, infection, coagulopathy, significant cardiac risk factors, or other medical risk factors for surgery
10. Pregnant and/or woman of childbearing age not using effective forms of birth control

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Mapping the limbic-associative STN in human using neuronal (single units & Local Field Potential (LFP)) responses to emotional stimuli during surgery and long term LFP recordings in PD and OCD patients | two years
  Mapping the limbic-associative STN in human using neuronal (single units & Local Field Potential (LFP)) responses to emotional stimuli during surgery and long term LFP recordings in Parkinson's diseae (PD) and Obsessive Compulsive Disorder (OCD) patients

CONTACTS AND LOCATIONS:
Overall Officials: Renana Eitan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel, Israel